CLINICAL TRIAL: NCT00291148
Title: A Comparative Single Center, Randomized Neuropathic Pain Assessment Study Involving Patients With Clinically Definite Multiple Sclerosis (MS) Receiving Treatment With Either Pregabalin or Paroxetine
Brief Title: Neuropathic Pain Assessment Comparing Pregabalin and Paroxetine in Management of MS-induced Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS_B2005:168
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2011-03

CONDITIONS: Neuropathic Pain; Multiple Sclerosis
Keywords: Neuropathic pain; Multiple Sclerosis; pregabalin; paroxetine
MeSH Terms: conditions — Neuralgia; Multiple Sclerosis | interventions — Paroxetine; Pregabalin

ARMS (2):
- Paroxetine (Active Comparator)
  Interventions: Drug: paroxetine
- pregabalin (Active Comparator)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: paroxetine
  Arms: Paroxetine
Drug: pregabalin
  Arms: pregabalin

SUMMARY:
This is a comparative drug trial involving patients with clinically definite Multiple Sclerosis and documented neuropathic pain. Patients will be randomized to receive treatment with either paroxetine or pregabalin. After dose titration, participants will complete various pain scale assessments at several points during the study in order to determine the effectiveness of their assigned pain medication.

DETAILED DESCRIPTION:
General Objective:

To determine the effectiveness of drug treatment in the management of MS-induced neuropathic pain.

Specific Objectives:

* Comparatively assess the effectiveness and safety profile of pregabalin (Lyrica) and paroxetine (Paxil) in managing MS-induced neuropathic pain.
* Comparatively assess the effectiveness of pregabalin (Lyrica) and paroxetine (Paxil) in improving the quality-of-life associated with MS-induced neuropathic pain.

Study Design:

A comparative single center, randomized, open-label study involving patients with multiple sclerosis (MS) - induced neuropathic pain receiving treatment with either pregabalin (Lyrica®) or paroxetine (Paxil®).

The study will run for approximately one year, requiring individual participants' involvement for 8 weeks.

Participant Selection:

Individuals with clinically definite MS presenting with symptoms of neuropathic pain (as determined by clinician) that express interest in the study will be screened for eligibility.

Inclusion Criteria:

* Patients presenting with symptoms of neuropathic pain as determined by clinician, with a minimum VAS pain score of 40mm as determined by a baseline score (0mm = no pain, 100mm = worst pain).
* Male and female patients between the ages of 18 and 65 years old.
* Clinically definite multiple sclerosis as defined by clinical history review, neurological examination and positive MRI.
* EDSS scores of < 6.0.
* No known hypersensitivity to the study medications.
* Negative serum pregnancy test for all female patients of childbearing age; not currently breastfeeding.
* Not currently treated with pregabalin, gabapentin, paroxetine or another SSRI.
* No previous treatment failures with pregabalin or paroxetine.
* Baseline creatinine clearance (Clcr) of > 50mL/min.
* No significant hepatic insufficiency.
* If on other pain medications, must be on stable dose for at least 6 months and other medications must not elicit significant drug-drug interactions with study medications.

Study Procedures:

After obtaining informed consent (Visit 1), participants undergo various assessments, including pain/quality-of-life analyses (SF-MPQ, SF-36, VAS), physical/neurological exam and a standard blood test. Based on above inclusion criteria, participants will be randomized to either Group A (paroxetine) or Group B (pregabalin). Participants will be provided with prescriptions for assigned study medications as well as dosing instructions. A pain diary consisting of a single VAS scale will be provided to the participants, which are to be completed daily upon waking and should be used to rate the individual's average pain over the last 24 hours. Dosages of study medications will be titrated slowly over 3 weeks to lower likelihood of adverse events. After the three week titration phase, participants will return to the clinic (Visit 2) for a follow-up. Pain/quality-of-life assessments (as at Visit 1) will be completed again at this visit. In addition, average pain scores will be determined from daily pain diaries. Adverse events will be discussed and individual tolerability will be assessed. At this point, it will be determined if the patient will be maintained at the target dosage or if the dosage will be lowered to accommodate patient tolerability. Participants will be maintained at determined maintenance dose for 5 weeks, after which they will return to the clinic (Visit 3) for a final follow-up assessment. Participants will complete final pain/quality-of-life assessments, as well as the "Patient-rated Global Impression of Change". Adverse events and average pain scores will be reviewed. At the conclusion of the 8-week treatment phase, participants will have the option of remaining on their current study medication or be tapered off.

ELIGIBILITY:
Inclusion Criteria:

* • Patients presenting with symptoms of neuropathic pain as determined by clinician, with a minimum VAS pain score of 40mm as determined by a baseline score (0mm = no pain, 100mm = worst pain).

  * Male and female patients between the ages of 18 and 65 years old.
  * Clinically definite multiple sclerosis as defined by clinical history review, neurological examination and positive MRI.
  * EDSS scores of < 6.0.
  * No known hypersensitivity to the study medications.
  * Negative serum pregnancy test for all female patients of childbearing age; not currently breastfeeding.
  * Not currently treated with pregabalin, gabapentin, paroxetine or another SSRI.
  * No previous treatment failures with pregabalin or paroxetine.
  * Baseline creatinine clearance (Clcr) of > 50mL/min.
  * No significant hepatic insufficiency.
  * If on other pain medications, must be on stable dose for at least 6 months and other medications must not elicit significant drug-drug interactions with study medications.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pain levels (as determined by weekly Visual Analogue Scale for pain) | 8 weeks

SECONDARY OUTCOMES:
Short-Form 36 health outcomes survey (SF-36) | 8 weeks
Short-form McGill Pain Questionnaire (SF MPQ) | 8 weeks
Patient-rated Global Impression of Change (PGIC) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Micheal P Namaka, PhD, Principal Investigator — University of Manitoba; Dana A Turcotte, BSc Pharm, Principal Investigator — University of Manitoba
Locations (1):
- Multiple Sclerosis Clinic, Health Sciences Centre, Winnipeg, Manitoba, Canada